CLINICAL TRIAL: NCT03076229
Title: A Randomized Control Trial of Relationship Education: Project Harmony
Brief Title: Relationship Education:Project Harmony
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCF MFRI
Record Dates: First submitted 2017-02-08; First posted 2017-03-10 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Healthy Marriage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Marriage: Treatment (Experimental): Intervention: Behavioral: Healthy Marriage Program
  Interventions: Behavioral: Healthy Marriage Program
- Healthy Marriage: Wait-list Control (Experimental): Intervention: Behavioral: Healthy Marriage Program
  Interventions: Behavioral: Healthy Marriage Program

INTERVENTIONS:
Behavioral: Healthy Marriage Program — Provide the following allowable activities 1) marriage and relationship education/skills, 2) relationship enhancement, 3) premarital education, and 4) divorce reduction.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of relationship education (RE) for individuals and couples participating in Project Harmony.

DETAILED DESCRIPTION:
Although considerable research supports the positive effects of relationship education (RE) on relationship satisfaction and communication skills, the majority of existing research designs have favored pre/post or quasi-experimental designs. Furthermore, gaps in the empirical bases for RE remain regarding programmatic moderators that influence change. Consequently, there has been less emphasis on understanding which program elements contribute to positive change within couple relationships. To this end, Project Harmony seeks to conduct an impact local evaluation design utilizing a randomized control trial (RCT) to assess the effectiveness of relationship education between low income, ethnically diverse individuals and couples in the treatment group compared to the wait-list control group. Secondary research questions are focused on investigating mechanisms and moderators of change for the target population. Participants (individuals and couples) in Project Harmony will be randomly assigned to either the treatment or wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals and couples who are at least 18 years of age.

Exclusion Criteria:

* Does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
1200 participants with relational and interpersonal stressors | 6 months
  The primary research question for the proposed investigation is: What are the effects of relationship education on relationship satisfaction (as measured by the Dyadic Adjustment Scale); between participants who received the intervention (treatment group) as compared with participants who did not immediately receive the intervention (wait-list control group)?

SECONDARY OUTCOMES:
1200 participants with relational and interpersonal stressors | 6 months
  What are the effects of relationship education on dyadic coping (as measured by the Dyadic Coping Inventory); between participants who received the intervention (treatment group) as compared with participants who did not immediately receive the intervention (wait-list control group)?

OTHER OUTCOMES:
1200 participants with relational and interpersonal stressors | 6 months
  What are the effects of relationship education on communication (as measured by Communication Patterns Questionnaire-Short Form); between participants who received the intervention (treatment group) as compared with participants who did not immediately receive the intervention (wait-list control group)?

CONTACTS AND LOCATIONS:
Overall Officials: Sejal M Barden, PhD, Principal Investigator — University of Central Florida; Bridgette Toussaint, MS, Study Director — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No